CLINICAL TRIAL: NCT06671548
Title: A Phase 3 Multicenter, Randomized, Double-Blind, Placebo-Controlled, Parallel-Designed Efficacy and Safety Study to Evaluate Relugolix Tablets in Women With Heavy Menstrual Bleeding Associated With Uterine Fibroids
Brief Title: Efficacy & Safety Study of Relugolix in Women With Heavy Menstrual Bleeding Associated With Uterine Fibroids
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Qilu Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: QLG1079-301
Record Dates: First submitted 2024-11-01; First posted 2024-11-04 (Actual); Last update posted 2026-02-02 (Actual); Status verified 2026-01

CONDITIONS: Heavy Menstrual Bleeding; Uterine Fibroids
MeSH Terms: conditions — Menorrhagia; Leiomyoma | interventions — relugolix; Megestrol Acetate; Medroxyprogesterone Acetate

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Relugolix plus megestrol acetate/medroxyprogesterone acetate (the treatment group) (Experimental): Relugolix 40 mg co-administered with megestrol acetate 1 mg and medroxyprogesterone acetate 2 mg for 12 weeks followed by 12 weeks of daily oral relugolix 40 mg co-administered with megestrol acetate 1 mg and medroxyprogesterone acetate 2 mg..
  Interventions: Drug: Relugolix
- Placebo (the placebo group) (Placebo Comparator): Relugolix 40 mg placebo co-administered with megestrol acetate 1 mg placebo and medroxyprogesterone acetate 2 mg placebo for 12 weeks followed by 12 weeks of daily oral relugolix 40 mg co-administered with megestrol acetate 1 mg and medroxyprogesterone acetate 2 mg.
  Interventions: Drug: Relugolix placebo

INTERVENTIONS:
Drug: Relugolix — * Relugolix (40 mg) tablet administered orally once daily；
  * megestrol acetate (1 mg) administered orally once daily；
  * medroxyprogesterone acetate (2 mg) administered orally once daily
  Other Names: megestrol acetate; medroxyprogesterone acetate
  Arms: Relugolix plus megestrol acetate/medroxyprogesterone acetate (the treatment group)
Drug: Relugolix placebo — Relugolix (0 mg) tablet administered orally once daily and manufactured to match the relugolix tablet in size, shape, color, and odor.
  megestrol acetate (0 mg) administered orally once daily and manufactured to match the relugolix tablet in size, shape, color, and odor.
  medroxyprogesterone acetate (0 mg) administered orally once daily and manufactured to match the relugolix tablet in size, shape, color, and odor.
  Other Names: megestrol acetate placebo; medroxyprogesterone acetate placebo
  Arms: Placebo (the placebo group)

SUMMARY:
The goal of this clinical trial is to determine the benefit of relugolix 40 milligrams (mg) once a day compared with placebo in heavy menstrual bleeding associated with uterine fibroids. The main question[s] it aims to answer are:

* the benefit of relugolix 40 mg once daily in women with heavy menstrual bleeding associated with uterine fibroids
* the safety of relugolix 40 mg once daily in women with heavy menstrual bleeding associated with uterine fibroids

DETAILED DESCRIPTION:
This study is a phase 3 multicenter, randomized, double-blind, placebo-controlled, parallel-designed efficacy and safety study to evaluate 12 weeks of oral daily relugolix 40 mg co-administered with megestrol acetate 1 mg and medroxyprogesterone acetate 2 mg (the treatment group) or 12 weeks of daily oral relugolix 40 mg placebo (the placebo group) followed by 12 weeks of daily oral relugolix 40 mg co-administered with megestrol acetate 1 mg and medroxyprogesterone acetate 2 mg.

Approximately 120 women with heavy menstrual bleeding associated with uterine fibroids will be enrolled and randomized 2:1 to the treatment group (N=80) or placebo group (N=40).

Stratification variables will include mean screening menstrual blood loss volume (< 225 mL versus ≥ 225 mL) by the alkaline hematin method.

The study consists of a screening period (up to ~13 weeks), a double-blind treatment period (12 weeks), an open-label treatment period (12 weeks) and a follow-up period (4w).

Safety will be assessed throughout the study by monitoring adverse events, vital signs, physical examinations, clinical laboratory tests, 12-lead electrocardiograms, and assessments of bone mineral density.

ELIGIBILITY:
Inclusion Criteria:

* Premenopausal female aged 18 or older
* Diagnosis of uterine fibroids confirmed by transvaginal/rectal ultrasound during the screening period
* Heavy menstrual bleeding caused by uterine fibroids
* Breast ultrasound results during the screening period meet the BI-RADS classification of 1 to 3
* Able to understand and comply with the study procedures and methods, voluntarily participate in this trial, and sign the informed consent form in writing

Exclusion Criteria:

* History of bilateral oophorectomy, or planned to undergo hysterectomy, bilateral oophorectomy, or other surgical procedures during the study period.
* Previous treatment with gonadotropin-releasing hormone (GnRH) agonists or GnRH antagonists for uterine fibroids has failed.
* History of or current osteoporosis or other metabolic bone disease.
* History of malignant tumor within 5 years prior to screening, except for cured skin cancer, basal cell carcinoma, and other localized malignant tumors.
* History of drug abuse, alcohol abuse, or drug dependence within 2 years prior to screening.
* Presence of an in situ copper intrauterine device (IUD) or a progestin-containing IUD implant/subdermal contraceptive implant during the screening period; subjects who can remove the IUD/subdermal contraceptive implant at least 1 month before enrollment may be allowed to participate.
* Baseline bone mineral density Z-score of < -2.0 at the lumbar spine, total hip, or femoral neck during the screening period.
* Any other factors that the investigator deems unsuitable for participation in this trial.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2024-01-15 (Actual); Primary Completion 2026-11-12 (Estimated); Study Completion 2027-01-07 (Estimated)

PRIMARY OUTCOMES:
Percentage Of Participants Who Achieved A Menstrual Blood Loss (MBL) Volume Of < 80 mL And ≥ 50% Reduction From Baseline MBL Volume | From Baseline up to the last 35 days of the double-blind treatment period
  A responder was a participant who had MBL volume of < 80 mL and at least a 50% reduction from baseline MBL volume over the last 35 days of the double-blind treatment period. All returned feminine products collected at each clinical visit were analyzed by the alkaline hematin method to obtain the MBL volume. MBL volume was measured over the Week 12/early termination feminine product collection interval (up to 35 days prior to the last dose of double-blind treatment). The percentage of participants who were responders are presented.
  As per the objective of the study, the pre-specified primary efficacy analyses compared relugolix plus megestrol acetate 1 mg and medroxyprogesterone acetate 2 mg with placebo. Therefore, only relugolix plus megestrol acetate 1 mg and medroxyprogesterone acetate 2 mg and placebo arms are presented.

SECONDARY OUTCOMES:
Percentage Of Participants With Amenorrhea Over The Last 35 Days Of the double-blind treatment period | From Baseline up to the last 35 days of the double-blind treatment period
  Following the administration of the investigational product, amenorrhea was defined as the central laboratory-confirmed measurement of blood loss volume <5 mL (including no bleeding) over a continuous 56-day period using feminine products.
  As per the objective of the study, the pre-specified secondary efficacy analyses compared relugolix plus megestrol acetate 1 mg and medroxyprogesterone acetate 2 mg with placebo. Therefore, only relugolix plus megestrol acetate 1 mg and medroxyprogesterone acetate 2 mg and placebo arms are presented.

CONTACTS AND LOCATIONS:
Locations (1):
- Peking Union Medical College Hospital, Beijing, China